CLINICAL TRIAL: NCT00221858
Title: Regional Anesthesia Database
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Other Study IDs: UHN02-0508-E
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Regional Anesthesia

STUDY DESIGN:
Time Perspective: Other

INTERVENTIONS:
Procedure: Ultrasound guided blocks

SUMMARY:
This is a quality assurance database to prospectively examine regional anesthesia outcomes at Toronto Western Hospital.

ELIGIBILITY:
Inclusion Criteria:Patients having regional anesthesia -

Exclusion Criteria:Patients not having regional anesthesia

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-08 (Actual); Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent WS Chan, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada